CLINICAL TRIAL: NCT01163162
Title: The Effect of Paricalcitol on Creatinine Filtration, Secretion and Glomerular Filtration Rate
Acronym: Paricalcitol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1003-15
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Vitamin D
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paricalcitol (Experimental): After baseline measurements are complete, pt will receive 2 mcg Paricalcitol (Zemplar) for 7 consecutive days. After this, Kidney function will again be measured. The pt will then be washed off the paricalcitol for 7 days then kidney function will be measured for the last time.
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Paricalcitol — 2 mcg oral Paricalcitol once per day for 7 days
  Other Names: Zemplar

SUMMARY:
The purpose of this study is to study the effects of Paricalcitol (Zemplar) on kidney functioning. The investigators hypothesize that the increase in serum creatinine observed in recent paricalcitol trials is a function of reduced creatinine secretion and not an actual reduction in kidney function. 16 patients will have kidney function measured via iothalamate clearance at baseline, after 7 days of paricalcitol treatment and after 7 days of being washed off the paricalcitol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Stage 3 or 4 CKD
* Ability to give informed consent

Exclusion Criteria:

* Serum Calcium > 10 g/dL
* Serum Phosphorous > 6 g/dL
* On > 400 units/d Vitamin D therapy
* Receiving cimetidine, triamterene, or trimethoprim, drugs that block creatinine secretion
* On vitamin D receptor activators (paricalcitol, calcitriol or Zemplar)
* Allergic to radiocontrast dye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Agarwal, MD, Principal Investigator — Indiana University
Locations (1):
- Roudebush VA Medical Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Agarwal R, Hynson JE, Hecht TJ, Light RP, Sinha AD. Short-term vitamin D receptor activation increases serum creatinine due to increased production with no effect on the glomerular filtration rate. Kidney Int. 2011 Nov;80(10):1073-9. doi: 10.1038/ki.2011.207. Epub 2011 Jun 29. PMID 21716260

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paricalcitol
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Paricalcitol
Number analyzed (Participants) | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 69.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Secondary Outcome: Creatinine Clearance
Description: The primary outcome variable will be creatinine clearance. Subject will be used as random variable and maximal likelihood estimation methods will be used. We expect no differences between periods.
Time Frame: 1 Week
Measure: Mean (95% Confidence Interval); unit: ml/min
Arm/Group | Paricalcitol
Number analyzed (Participants) | 16
ml/min | 0.49 [-0.26 to 1.23]

2. Secondary Outcome: Serum Creatinine
Description: We expect serum creatinine to confirm the results of creatinine clearance.
Time Frame: 1 Week
Measure: Mean (95% Confidence Interval); unit: mg/dl/day
Arm/Group | Paricalcitol
Number analyzed (Participants) | 16
mg/dl/day | 0.010 [0.001 to 0.019]

3. Primary Outcome: 24-hour Urine Creatinine Excretion Rate
Description: We expect the 24 hour urine creatinine excretion rate to show no differences between groups.
Time Frame: 1 Week
Measure: Mean (95% Confidence Interval); unit: mg/24hour/day
Arm/Group | Paricalcitol
Number analyzed (Participants) | 16
mg/24hour/day | 17.6 [0.5 to 34.6]

ADVERSE EVENTS:
Arm/Group | Paricalcitol
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paricalcitol (N=16)
Dizziness (General disorders) | 2 (2)
Skin irritation (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes